CLINICAL TRIAL: NCT05296980
Title: Validation of a Multidomain Neuropsychological Intervention for Individuals at Risk of Dementia: the REMINDER Program
Brief Title: Validation of the REMINDER Dementia Risk Reduction Program
Acronym: REMINDER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Ana Rita Silva, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: REMINDER
Record Dates: First submitted 2022-02-22; First posted 2022-03-25 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Healthy Aging; Risk Reduction; Old Age; Dementia
MeSH Terms: conditions — Risk Reduction Behavior; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- REMINDER program online (Experimental): The REMINDER program in this arm will be delivered by videoconferencing. It will integrate 20 sessions (with approximate length of 45-60 min), therapist-mediated, carried out twice a week, over a period of 12 weeks. Psychoeducation sessions and part of the reminiscence and memory strategies training sessions will be facilitated in groups, as means to promote social support and modeling, and the remaining will be individual sessions. Several activities aimed to promote personal development and definition and achievement of meaningful goals will be included in the program, and the program will be manualized to facilitate its future dissemination and implementation
  Interventions: Behavioral: REMINDER
- REMINDER program face-to-face (Experimental): The REMINDER program in this arm will be delivered face to face. It will integrate 20 sessions (with approximate length of 45-60 min), therapist-mediated, carried out twice a week, over a period of 12 weeks. Psychoeducation sessions and part of the reminiscence and memory strategies training sessions will be facilitated in groups, as means to promote social support and modeling, and the remaining will be individual sessions. Several activities aimed to promote personal development and definition and achievement of meaningful goals will be included in the program, and the program will be manualized to facilitate its future dissemination and implementation
  Interventions: Behavioral: REMINDER
- Brain psychoeducation program (Sham Comparator): The control condition will have the same length as the experimental harms, including 20 psychoeducation sessions, with information regarding dementia modifiable risk factors, information on healthy lifestyles, and brain health promotion.
  Interventions: Behavioral: Brain health Psychoeducation

INTERVENTIONS:
Behavioral: REMINDER — The REMINDER program is a therapist-mediated manualized neuropsychological intervention, involving training skills to stimulate cognitive reserve, socialization and personal development, to diminish the risk of cognitive decline.
  Arms: REMINDER program face-to-face; REMINDER program online
Behavioral: Brain health Psychoeducation — Delivery of psychoeducation sessions about dementia modifiable risk factors, brain health solutions and lifestyle change tips.
  Arms: Brain psychoeducation program

SUMMARY:
Until now, neuropsychological interventions aimed to optimize cognitive function and to have functional impact in individuals at risk of AD (MCI patients) were scarce in validity studies. While some RCTs have been developed in cognitive training interventions, comparative studies of merged interventions (cognitive, social and behavioral stimulation) with adequate control groups are absent, diminishing the professionals' trust on the adoption of these interventions for supporting patients. As such, the present proposal will develop a validation trial testing a multicomponent neuropsychological intervention (REMINDER), based on personal development, cognitive compensatory aids, meaningful goals setting, and behavior change techniques. The investigators will analyze its short/long-term gains and AD conversion rates. By aiming to provide a good validation study for REMINDER, the investigators will examine neurobiological, neurocognitive and functional outcomes of this intervention in comparison with an active control group (psychoeducation) in order to foster an effective outcome assessment of an intervention for individuals at risk of AD.

DETAILED DESCRIPTION:
The overarching tenet of this project is that, by providing a manualized multidomain intervention - REMINDER - that engages at risk individuals in the aims of this protocol, it can have a significant impact on health outcomes, optimizing healthier lifestyles and these being also understood along with the neurodegeneration signs of this impact.

The specific aims of this study will be:

* Recruit community-dwelling individuals with increased risk of dementia using CAIDE dementia risk score (with APOE, when available).
* Evaluate the REMINDER program (in comparison to an active control group (CT) - psychoeducation sessions) immediate effects regarding global cognition and functionality (primary outcomes) and neuropsychological, biochemical and neuroimaging outcomes (secondary outcomes).
* Determine the persistence of effects and begin characterizing the temporal course of putative benefits at 6-, and 18-months follow-up.
* Investigate the role of biomarkers (imaging and biochemical) in explaining the response to intervention and persistence of the effects and its correlation with neuropsychological and functionality measures.
* Measure the conversion rates from MCI to AD between the REMINDER and active control groups (at 24- months follow-up).

Our ultimate goal is to make available a scientifically validated and scalable intervention that helps prevent dementia in older adults at risk. By confirming the efficacy of REMINDER to prevent cognitive impairment and concluding for its medium-term efficacy to improve global cognitive function and healthy life habits the investigators are contributing to one of the WHO goals (Goal 3 - ensure healthy lives and promote well-being for all at all ages) by addressing risk reduction and management of a global health risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older
* CAIDE dementia risk score >8
* Cognitive function: absence of significant cognitive impairment as per the Addenbrooke's Cognitive Examination-REVISED
* Free of physical disabilities that preclude participation in the study
* Willing to complete all study-related activities for 12 weeks

Exclusion Criteria:

* Mild cognitive impairment or dementia;
* Presence of any neurological event in their medical history that could compromise actual cognition.
* Presence of any severe psychiatric disorder (mild depressive and anxiety symptoms meet inclusion criteria).
* Unability to travel to the site where the sessions will be delivered (if so randomization will be circumscribed between the experimental harm REMINDER online and the control group.
* Illiteracy

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Cognitive status composite | Post intervention (1 week after the intervention sessions completion)
  A composite score including the individual scores with Addenbrooke's Cognitive Examination - Revised (ACE-R) (0-100, higher scores meaning better outcome), that includes the Mini Mental State Examination - MMSE (0-30, with higher scores meaning better outcome), Subjective Cognitive Decline Questionnaire (SCDQ), Trail Making Test A and B (TMT A & B), Verbal Fluency - Phonemic (P, M and R) and Categories (Animals), Stroop Test, Free and Cued Selective Reminding Test (FCSRT) will be generated to work as primary outcome.
Functionality status | Post intervention (1 week after the intervention sessions completion)
  A composite score incorporating Adults and Older Adults Functional Assessment Inventory (IAFAI), University of California San Diego Performance-Based Skills Assessment (UPSA) will be used.
Blood biomarkers of neural damage | Post intervention (1 week after the intervention sessions completion)
  blood Neurofilament light chain (NfL) will be measured and tested as an outcome immediately after the intervention
Cognitive status composite | Follow - up (12 months after the intervention)
  A composite score including the individual scores with Addenbrooke's Cognitive Examination - Revised (ACE-R), that includes the Mini Mental State Examination - MMSE (screening tools to consider eligibility), Subjective Cognitive Decline Questionnaire (SCDQ), Trail Making Test A and B (TMT A & B), Verbal Fluency - Phonemic (P, M and R) and Categories (Animals), Stroop Test, Free and Cued Selective Reminding Test (FCSRT) will be generated to work as primary outcome
Functionality status | Follow - up (12 months after the intervention)
  A composite score incorporating Adults and Older Adults Functional Assessment Inventory (IAFAI), University of California San Diego Performance-Based Skills Assessment (UPSA) will be used.
Cognitive status composite | Follow - up (24 months after the intervention)
  A composite score including the individual scores with Addenbrooke's Cognitive Examination - Revised (ACE-R), that includes the Mini Mental State Examination - MMSE (screening tools to consider eligibility), Subjective Cognitive Decline Questionnaire (SCDQ), Trail Making Test A and B (TMT A & B), Verbal Fluency - Phonemic (P, M and R) and Categories (Animals), Stroop Test, Free and Cued Selective Reminding Test (FCSRT) will be generated to work as primary outcome
Functionality status | Follow - up (24 months after the intervention)
  A composite score incorporating Adults and Older Adults Functional Assessment Inventory (IAFAI), University of California San Diego Performance-Based Skills Assessment (UPSA) will be used.

SECONDARY OUTCOMES:
Brain changes | Post intervention (2 weeks after the intervention sessions completion)
  hippocampus volume and DMN connectivity will be measured pre and post intervention in the RCT phase
Mood status | Post intervention (1 week after the intervention sessions completion)
  The Geriatric Depression Scale Short Form (GDS-15) (0-15, with higher scores meaning worse outcomes) and and The Geriatric Anxiety Inventory- Short Form (GAI-SF, 0-5, with higher scores meaning worse outcome) scores will be measured
Mood status | Follow-up (12 months after the intervention)
  The Geriatric Depression Scale Short Form (GDS-15) (0-15, with higher scores meaning worse outcomes) and and The Geriatric Anxiety Inventory- Short Form (GAI-SF, 0-5, with higher scores meaning worse outcome) scores will be measured.
Perceived quality of life | Post intervention (1 week after the intervention sessions completion)
  A measure of quality of life - World Health Organization Quality of Life - Old WHOQOL-OLD)will be incorporated to examine the effects of the program in self perceptions of well being. Higher scores mean better outcome
Perceived quality of life | Follow-up (12 months after the intervention)
  A measure of quality of life - World Health Organization Quality of Life - Old WHOQOL-OLD)will be incorporated to examine the effects of the program in self perceptions of well being. Higher scores mean better outcome
Perceived Self Efficacy | Post intervention (1 week after the intervention sessions completion)
  A measure of self efficacy - Self Efficacy for Meaningful Activities (SEMActiv) will be implemented to examine self-efficacy, with higher scores meaning better outcome
Perceived Self Efficacy | Follow-up (12 months after the intervention)
  A measure of self efficacy - Self Efficacy for Meaningful Activities (SEMActiv) will be implemented to examine self-efficacy, with higher scores meaning better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psychology and Educational Sciences, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
Open science plans will involve the sharing of IPD with other researchers, clearly anonymized in order to promote the studies replication. We are still building our plan for data sharing and we will update as soon as it is defined.

REFERENCES:
- [Derived] Silva AR, Baptista C, Baldeiras I, Pinho MS, Lima M, Afonso RM. REMINDER program: a randomized controlled trial protocol of a neuropsychological intervention for lifestyle modification in older adults at risk of dementia. BMC Geriatr. 2025 Dec 10;26(1):48. doi: 10.1186/s12877-025-06714-x. PMID 41366742